CLINICAL TRIAL: NCT03224078
Title: Utilization and Trans-sectoral Patterns of Care for Patients Admitted to Emergency Departments in Germany
Brief Title: Emergency Department Utilization in Germany
Acronym: INDEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Zentralinstitut für die Kassenärztliche Versorgung in Deutschland (Unknown); University of Magdeburg (Other); Wissenschaftliches Institut der AOK (WIdO) (Unknown); Technische Universität Berlin (Other); Technologie- und Methodenplattform für die vernetzte medizinische Forschung (TMF) (Unknown); OFFIS - Institut für Informatik (Unknown)
Responsible Party: Principal Investigator, Martin Moeckel, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: EA4/086/17
Record Dates: First submitted 2017-06-23; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult Emergency Department Patients: adult patients that were treated with any condition in one of the participating emergency departments in 2016 (n≈680.000 cases)
  Interventions: Other: data extraction

INTERVENTIONS:
Other: data extraction — No Special interventions except from data extraction form the respective routine data sources are planned .

SUMMARY:
The overall aim of INDEED is to facilitate trans-sectoral and interdisciplinary health services research of emergency care in Germany.

Clinical hospital data from 15 to 20 emergency departments in Germany will be linked to routine ambulatory health care data provided by the Association of Statutory Health Insurance Physicians (Kassenärztliche Vereinigung, KV). INDEED will identify health care gaps and inadequate resource allocation as well as develop strategies for adaptations of the health care system to existing demands.

DETAILED DESCRIPTION:
B a c k g r o u n d:

Emergency departments nationally and internationally are challenged by a continuously increasing number and complexity of patients and consequent crowding. International studies showed that crowding is associated with unfavourable outcomes. Emergency departments are an important interface between the outpatient and inpatient health care sectors. Health care sectors in Germany are not organisationally cross-linked and data linkage for analysis of the health care system is not generally performed. Hence, there is a lack of data to trans-sectorally describe and monitor patients' pathways and patterns of care in the health care system.

RESEARCH AIMS:

The overall aim of INDEED is to facilitate trans-sectoral and interdisciplinary health services research of emergency care in Germany.

The primary objective of the project is to assess the trans-sectoral utilization of health care services of patients 2 years prior and 1 year after treatment in an emergency department. Patterns of adequate, inadequate and potentially avoidable care will be examined.

The secondary aim is to identify patient clusters with comparable needs of health care provision. Within clusters and for all patients combined INDEED will examine health care needs and gaps as well as factors that influence emergency department visits, disease progression, comorbidities and mortality.

METHODS:

Clinical hospital data from 15 to 20 emergency departments in Germany will be linked to routine ambulatory health care data provided by the Association of Statutory Health Insurance Physicians (Kassenärztliche Vereinigung, KV).

A secondary data analysis of linked routinely collected hospital information system and health insurance data of all adult patients that were treated with any condition in one of the participating emergency departments in 2016 (n≈680.000 cases) will be performed. Data analysis will cover the pattern of utilization of health care, identification of subgroups with comparable need of health care provision, of factors that influence emergency department visits and factors for ambulatory care sensitive conditions (ACSC) or inpatient treatment. Study results will be evaluated considering age, multimorbidity and gender aspects as well as the health system and health economic perspective. Thereby INDEED will identify health care gaps and inadequate resource allocation as well as develop strategies for adaptations of the health care system to existing demands.

ELIGIBILITY:
Inclusion Criteria:

* adult ED patients who attended one of the participating EDs in 2016
* patients with public health insurance

Exclusion Criteria:

* no exclusion criteria are applied

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with public health insurance who attended one of the participating EDs in 2016 will be included in this research Project.
Sampling Method: Non-Probability Sample
Enrollment: 680000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adequate, inadequate and avoidable ED-visits | Baseline
  Prevalence of adequate, inadequate and avoidable ED-visits will be operationalized by a) patients with low utilization of primary health care, b) low urgency, c) preventable conditions, d) chronic diseases that could have been adequately controlled, e) frequent-users, f) patients without contact to a physician in the ED ("left without being seen").

SECONDARY OUTCOMES:
Characterization of health care resource utilization before and after an ED-visit | from 2 years before until 1 year after ED-visit (2014-2017)
  Descriptive analysis of number of visits to primary care physicians before and after the ED visit. The utilization of primary health care will be assessed two years before and one year after the year of the ED visit. ED-visits will be analyzed for the year 2016, this outcome measure will be analyzed for the years 2014-2017.
influencing factors on avoidable ED-visits | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency.
influencing factors on adequate ED-visits | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency.
influencing factors on inadequate ED-visits | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency.
Exploratory analysis of influencing factors on increased health care costs. | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency. Outcome will be treatment costs in the ambulatory sector as well as in-hospital diagnosis related group (DRG) for hospitalized patients
Exploratory analysis of influencing factors on patient-related mortality | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency. Outcome measure: mortality two years after the year of the ED-visit.
Exploratory analysis of influencing factors on morbidity | from 2 years before until 1 year after ED-visit (2014-2017)
  influencing factors: sex, age, number of contacts to primary care physician, day and time of ED-admission, diagnoses, medication, admission mode, urgency. Outcome measure: morbidity two years after the year of the ED-visit.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Möckel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin - Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data could be made available to other researchers on reasonable request and if data protection requirements are met.